CLINICAL TRIAL: NCT01863303
Title: Epidemiological Study of Colorectal Cancer in WuHan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wuhan Pu-Ai Hospital (Other)
Collaborators: Wuhan University (Other); Hubei Cancer Hospital (Other); Huazhong University of Science and Technology (Other); Wuhan Iron and Steel Workers' Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R201206DCAPC
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Diarrhea; Constipation; Melena; Neoplasm; Colonic Neoplasms; Pain
Keywords: colorectal cancer; epidemiology; industry; genetic
MeSH Terms: conditions — Diarrhea; Constipation; Melena; Neoplasms; Colonic Neoplasms; Pain; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample or neoplasm from high risk group
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The incidence risk of colorectal cancer （CRC） is increasing at 4.2% year by year in China. Most effective way to reduce the death rate of CRC patients is to diagnose in quite an early stage. QiaoKou District is a chemical industry Zone of Wuhan with a long history, which has few data of CRC epidemiology. The investigators design the primary CRC screening for this district by healthy questionnaire, Fecal Occult Blood Test(FOBT) and colonoscopy. HanYang Areo has been chosen as Control for its non-industry environment.The crowd would be screen biennially. The high risk group would be intervened, such as resection of polyps or other specific treatment. A follow-up registration database has been built for analysis the relationship between incidence or death rate to high risk factors, such as age, life environment, lifestyles, base diseases and family history of cancer.

This study will provide some epidemiology dates of CRC to the local Government, and assist the governor to built a more effective screening system of CRC.

DETAILED DESCRIPTION:
For this study, you will be asked to complete a personal interview. During the interview, you will be asked questions about your demographics (age, sex, etc.), underlying diseases, lifestyle, family history of cancer, awareness of CRC. It should take around 30 minutes to complete the interview.

Residents in high risk group need to have some special tests, including FOBT and colonoscopy. Intestinal neoplasm will be suggested to biopsy or remove under colonoscopy for pathological examination. All tests are free. The interviews will be performed in Residential area and special tests will be done in the hospital during a regularly scheduled visit to Pu-Ai hospita.You may be contacted at home by phone so that researchers can collect information about any changes in your health status.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 40-74
2. Resident of Qiaokou Areo，and at least ten years living history in this district
3. Willing and able to provide written informed consent and authorization
4. Willing to a personal interview and have some special tests

Exclusion Criteria:

1. Under 43 or older than 74 years of age
2. History of colorectal cancer
3. Mental disorders

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coulp of this study from a chemical industry Zone of Wuhan with a long history,seriously polluted environment， which has few data of CRC epidemiology.
  HanYang Areo has been choosen as Control for its non-industry environment
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2012-06; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
incidence of CRC | June 2022 (up to 10 years)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Li, doctor, Study Director — Zhongnan hospital of Wuhan university, China